CLINICAL TRIAL: NCT06446089
Title: The Feasibility of a Culturally Tailored Mobile App-based Thinking Healthy Program for Mental Health Support of East Asian Pregnant Immigrants in Canada
Brief Title: A Chinese Version of the Thinking Health Program for East Asian Pregnant Immigrant People in Canada
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Shahirose Sadrudin Premji, Professor and Sally Smith Chair in Nursing, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6041350; FRN 154988 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-05-23; First posted 2024-06-06 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Perinatal Depression
Keywords: immigrant women; East-Asian immigrants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adapted THP group (Experimental): Participants will be invited to complete three modules relevant to the health and well-being of mothers and fetus/infants during the perinatal period, through an Android based app on their mobile device.
  In addition, each section incorporates the three healthy thinking steps to help the mother negotiate each of the three areas.
  After the introductory session, each session involves four tasks that mothers are required to complete. The tasks include 1) a review of the key message from the previous section, 2) a review of the mood chart, 3) engaging in the three steps to thinking healthy on the designated area for the section, and 4) practicing suggested activities between sessions.
  Interventions: Behavioral: THP: cognitive behavior therapy and behavioral activation

INTERVENTIONS:
Behavioral: THP: cognitive behavior therapy and behavioral activation — The adapted THP takes into account cultural and linguistic characteristics of the participants. Participants will be invited to complete three modules on an Android based app on their mobile, populated with information and activities from the adapted THP.

SUMMARY:
The goal of this study is to determine the feasibility of using a psychosocial intervention culturally adapted in China to support perinatal mental well-being of Chinese immigrant pregnant women in Canada. The intervention is adapted from the Thinking Healthy Program (THP), available through a mobile application, and will be offered to Chinese immigrant pregnant women (22 weeks' gestation or greater) residing in Canada, who are over the age of 18, and speak Mandarin. The main questions this study aims to answer are:

* Will the Chinese version of the THP be acceptable to Chinese immigrant pregnant women residing in Canada and will they use the program which is delivered through a mobile App?
* How well does the process of recruiting, keeping participants in the study and helping them complete the activities work, so it can be used for a future larger study?

Women interested in the study and who meet the study criteria will complete a questionnaire at the start of the study, then use the THP for three weeks, complete questionnaires 3-4 weeks after completing the intervention and 6-8 weeks after having their baby(ies). Some may be asked to participate in an individual interview.

DETAILED DESCRIPTION:
Common mental health conditions during pregnancy include depression and anxiety. Having an immigrant status and belonging to an ethnic minority group is linked to an increased likelihood of perinatal mental health problems. The lack of culturally tailored and innovative intervention is a predominant factor affecting mental health outcomes for immigrant women. Psychological and psychosocial interventions have been reported to significantly improve non-migrant women's mental health. The Thinking Healthy Program (THP), a low-intensity, low-cost, psychosocial intervention ("talking therapies") based on cognitive behavioural therapy, is comprised of 12, 1-hour sessions with content organized in modules (e.g., preparing for the baby, baby's arrival) that have associated activities (e.g., mood chart). In China, the THP has been culturally and linguistically adapted using rigorous processes and delivered to support women in the management of perinatal depression. To improve access and ensure a more impactful outcome to the culturally adapted THP, a mobile App was created in China with a brief Chinese version of the culturally adapted THP.

The primary objective of this study is to (1) assess the feasibility (acceptability and usability) of the linguistically and culturally adapted THP delivered through a mobile App to Chinese immigrant pregnant women residing in Canada; and (2) examine the process of recruitment, retention, and adherence to intervention to inform a future trial. The secondary objective is to produce preliminary evidence on the effectiveness of the brief Chinese version of THP on immigrant women's mental well-being, specifically depression.

A sequential explanatory mixed-method feasibility study involving a pre-post design in which a single group will be assembled and assessed quantitatively at baseline, 3-4 weeks after initiation of brief Chinese version of the THP intervention and again at 6-8 weeks following the birth of their baby. A subset of participants that have engaged with the intervention (n=up to 15) will be invited to individual semi-structured telephone interview to share their experience with the intervention.

A convenience sample of 50 participants will be recruited for the intervention, with a subset of 15 participants to be individually interviewed via the telephone.

Participants will be recruited through social media (WeChat and Xiaohongshu), research team members' University mailing list, dissemination to professional colleagues (e.g., Obstetrics and Gynecologists), and collaboration with social and health-based organizations that serve the East Asian community in Canada.

At baseline, the sociodemographic characteristics, immigrant characteristics, health/obstetric history, and history of psychological well-being will be assessed. Potential covariates that will be assessed once include acculturation (baseline; Vancouver Index of Acculturation) and preterm birth (at 6 to 8 weeks postpartum) while all others including pregnancy-related anxiety (Pregnancy-Related Anxiety Scale), depression severity (Patient Health Questionnaire-9), somatic symptoms (Patient Health Questionnaire-15), psychological stress (Perceived Stress Scale-10), resilience (Connor-Davidson Resilience Scale-10), social support (Multidimensional Scale of Perceived Social Support), mother-infant relationship (prenatal section of the Pre- and Postnatal Bonding Scale), and patient activation (Behavioural Activation for Depression Scale) will be assessed at baseline and follow-up (3-4 weeks after initiation of intervention and/or 6 to 8 weeks post-partum), using the scales and instruments listed above.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at ≥ 22 weeks of gestation; AND
* ≥ 18 years old; AND
* are first or second-generation Chinese immigrants residing in Canada (who identify as someone with East Asian cultural and ethnic background born outside of Canada or have at least one parent born outside of Canada); AND
* understand both spoken and written Mandarin language; AND
* have access to internet and a smartphone with Android operating system or willing to download an Android emulator to operate the App; AND
* are willing to download and use the study mobile App with brief Chinese version of THP for "talking therapy" with accompanying activities.

Exclusion Criteria:

* Women currently being treated for mental conditions, including depression

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Score on the System Usability Scale (SUS) 10 points | 3-4 weeks after initiation of intervention
  Objective measurement of usability of internet-based cognitive behavioural therapy
Acceptability of app-based THP | 3-4 weeks after initiation of intervention
  Structured questions based on seven domains of Sekhon's Theoretical Framework of Acceptability
Recruitment to study | During recruitment to study, expected 4 months
  Through RedCap-captured data and study intervention App-derived user data. Number of participants approached and recruited to the study will be tracked, and reported in a participant flow diagram.
Retention in study | Through study completion, an average of 12 months.
  Number of participants lost to follow-up (i.e., these may include dropouts who use the brief Chinese version of the THP mobile App but fail to complete the follow-up assessments), as well as number of participants with partial or complete data for analysis will be tracked.
Adherence to intervention | Through intervention duration, an average of 3-4 weeks.
  Defined as the extent to which individuals experience the content of the brief Chinese version of the THP mobile App (i.e., average amount of time participants spend on the modules, average amount of time participants use of the health assistants and tools within the app). Measured through App-derived user data.

SECONDARY OUTCOMES:
Effectiveness of app-based THP | Baseline, 3-4 weeks after initiation of intervention, and 6-8 weeks post-partum
  Edinburgh Postnatal depression scale (EPDS; 10 items). Assess change of mean scores from baseline to treatment completion (at 3-4 weeks), and 6-8 weeks after the birth of the baby, adjusting for significant predictors (e.g. social support, mother-infant bonding).

OTHER OUTCOMES:
Pregnancy-related anxiety | Baseline, & 3-4 weeks after initiation of intervention
  Pregnancy-Related Anxiety Scale (10 items)
Somatic symptoms | Baseline, 3-4 weeks after initiation of intervention, and 6-8 weeks post-partum
  PHQ-15 (14 items)
Psychological stress | Baseline, 3-4 weeks after initiation of intervention, and 6-8 weeks post-partum
  Perceived Stress Scale (10 items)
Resilience | Baseline, 3-4 weeks after initiation of intervention, and 6-8 weeks post-partum
  Connor-Davidson Resilience Scale (10 items)
Social support | Baseline, 3-4 weeks after initiation of intervention, and 6-8 weeks post-partum
  Multidimensional Scale of Perceived Social Support (12 items)
Mother-infant relationship | Baseline, 3-4 weeks after initiation of intervention, and 6-8 weeks post-partum
  Pre- and Postnatal Bonding Scale (5 items)
Patient activation | Baseline & 3-4 weeks after initiation of intervention
  PREMIUM Abbreviated activation scale (5 items)
Preterm birth | 6-8 weeks post-partum
  Pregnancy/Delivery/Puerperium Outcome questions (5 items)
Acculturation | Baseline
  Vancouver Index of Acculturation (18 items)
Depression severity | Baseline, 3-4 weeks after initiation of intervention, and 6-8 weeks post-partum
  Patient Health Questionnaire-9 (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Shahirose Premji, PhD, NP, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No